CLINICAL TRIAL: NCT07009405
Title: Continuous Monitoring of Intravenous Site Events With a Wireless Thermal Measurement Device During Outpatient Infusion Procedures
Brief Title: Assessment Intravenous Site Events During Outpatient Infusion Procedures With a Wireless Thermal Measurement Device During
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhaeos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2025-02
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: IV Infiltration; IV Extravasation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- IV Infusion Patients (Experimental): Pediatric patients over the age of 12 and adult patients with planned outpatient infusion procedures scheduled will be enrolled in this study.
  Interventions: Device: non-invasive thermal infusion site monitoring NTISM device

INTERVENTIONS:
Device: non-invasive thermal infusion site monitoring NTISM device — Non-invasive thermal infusion site monitoring NTISM device for detecting extravasation and infiltration events using thermal anisotropy measurements

SUMMARY:
This study evaluates a Non-invasive Thermal Infusion Site Monitor (NTISM) device when used during routine outpatient infusion treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to receive an infusion therapy of at least 30 minutes in length
2. Region of intact skin proximal to the infusion catheter insertion site that is appropriate in size for application of the study device
3. Signed informed consent
4. Available for 15 minutes of post-measurement monitoring following removal of the study device

Exclusion Criteria:

1. Patient is under 12 years of age
2. Patient-reported history of serious adverse skin reactions to silicone-based adhesives or Tegaderm
3. Use of the study device would interfere with standard patient care that cannot be delayed, or participation in the study will interfere with, or be detrimental to, administration of optimal healthcare to the subject
4. Investigator judges that the intravenous

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Thermal skin measurements | Up to 12 hours of monitoring with a 15-minute follow-up period.
  Exploratory assessment of thermal skin measurements taken with the study device

CONTACTS AND LOCATIONS:
Overall Officials: R. Chad Webb, Principal Investigator — Rhaeos, Inc.
Locations (1):
- Infusacare, Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: No